CLINICAL TRIAL: NCT04970615
Title: Educating Brain Tumor Patients Using Patient-specific Actual-size Three-dimensional Printed Models: a Case-control Study
Brief Title: Educating Brain Tumor Patients Using Patient-specific Actual-size Three-dimensional Printed Models
Acronym: IMAGE-3D
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sümeyye Sezer (Other)
Responsible Party: Sponsor-Investigator, Sümeyye Sezer, MD, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Other Study IDs: 2021-7292
Record Dates: First submitted 2021-06-15; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Brain Tumor; Glioma; Glioblastoma; Astrocytoma; Neoplasm, Brain; Oligodendroglioma; Patient Education as Topic; Decision Making, Shared
Keywords: brain tumor; glioma; three-dimensional printing; patient education; three-dimensional model
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma; Astrocytoma; Oligodendroglioma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Two-dimensional images: Patients who receive pre-operativeinformation while the two-dimensional MR images are being shown to them by the neurosurgeon.
- Three-dimensional printed model: Patients who receive pre-operative information while the three-dimensional printed models are being shown to them by the neurosurgeon.
  Interventions: Device: Three-dimensional printed model

INTERVENTIONS:
Device: Three-dimensional printed model — Three-dimensional printers are able to print physical objects in real size and colours. As a respresentative of the real tumor, a personalized three-dimensional model enables visualization of the patient-specific tumor and eloquent areas.
  Groups: Three-dimensional printed model

SUMMARY:
Patient education plays an essential role in patient-centered care as it enhances patient satisfaction and information comprehension. However, about 40-80% of the information patients receive from healthcare professionals is forgotten and about half of the information patients remember is incorrect. To give informed consent, patients must be able to understand and recall the discussed information correctly. This is especially important in brain tumor patients, in which different treatment options determine outcome and risks. The goal of treatment in brain tumors is resection as completely as possible, without damaging healthy brain tissue. To this end, patients must understand the complex relation of the tumor to healthy brain tissue. This relation is different in each patient and three-dimensional (3D) in nature. Current two-dimensional visual tools lack the ability to properly display these complex 3D relations. In this study, we will investigate the effect of the use of 3D models in patient education, taking into account patient specific factors that might act as confounders. We will conduct a case control, multi-center study in the Radboud University Medical Center (Radboudumc) Maastricht University Medical Center (MUMC). Patients will be enrolled in the control group until inclusion for the control group is completed (n=30), after which patients will be enrolled in the intervention group (n=30). Patients will be cognitively tested using the Amsterdam Cognition Scale (ACS). After the consultation with their neurosurgeon, patients will be asked to fill out two questionnaires, consisting of two parts (patient experiences and information recall), one week apart.

DETAILED DESCRIPTION:
Objectives The main goal of this project is to evaluate the role of 3D models on different aspects of patient education (patient experiences and information recall) in patients with brain tumors by comparing these to the use of standard 2D Magnetic Resonance (MR) images. A secondary goal is to gain more insight into the experiences of the close ones of the patients.

Study population We will conduct a case control, multi-center study in the Radboud University Medical Center (Radboudumc) Maastricht University Medical Center (MUMC). Patients will be enrolled in the control group until inclusion for the control group is completed (n=30), after which patients will be enrolled in the intervention group (n=30). The control group will consist of patients who will be informed using MR images during pre-operative consultations. The intervention group will be informed using personalized, life-size 3D models during pre-operative consultations. Inclusion time is estimated to be around 2 years.

Sample size Previous studies on this topic are scarce. In our experimental study on this subject [Sezer et al. 2020], we found an improvement of 5% (minimum expected difference, D) in information recall when using 3D models compared to 2D models. The standard deviation (SD) for information recall based on this study is approximately 5. With a significance criterion of 0.05 and power of 0.90 we calculated a total sample size of 42. For this study, however, we expect to find a smaller effect size due to the confounding factors (cognitive functioning, emotional status) which were eliminated in our experimental study in healthy individuals. Therefore we want to enroll 30 patients in each group (total sample size 60).

Study procedures Eligible patients will be asked to participate by their clinician or nurse practitioner who will they will receive an information letter and informed consent (attachment E1.1). The researcher will contact the patient to officially collect the informed consent form. Afterwards, the researcher will send out the link to the questionnaires collecting the baseline characteristics, emotional status questionnaire (HADS) and the ACS. The patient will be instructed to finish these questionnaires before the pre-operative consultation. Pre-operative preparation will be the same for the control and intervention group. The only difference will be the visual tool used in the pre-operative consult. Afterwards, the patient will be called by the researcher on the same or following day. A link will be sent out with the questionnaires on experiences, information recall and chosen treatment for the brain tumor. All questionnaires will be collected through Castor EDC © 2019.

The clinician will also be asked to fill out the questionnaire on information recall.

After the pre-operative consultation, we will ask the participant whether we can contact their close one. After reading the information letter and signing the informed consent the close one will receive the online questionnaires testing information recall and experiences. Both questionnaires will be collected through Castor EDC © 2019.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a brain tumor
* functional imaging (MRI, functional MRI (fMRI) and Diffusion Tensor Imaging (DTI)) requested for pre-operative planning

Exclusion Criteria:

* Inadequate understanding of the Dutch language
* Inability to independently use a computer

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a brain tumor who undergo functional imaging (MRI, functional MRI (fMRI) and Diffusion Tensor Imaging (DTI)) requested for pre-operative planning after which they undergo a pre-operative consultation.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Immediate information recall | 24 hours
Delayed information recall | One week
Patient experiences | 24 hours

SECONDARY OUTCOMES:
Inclusion rate of patients meeting the inclusion criteria | 30 months
Number of patients with completed follow-up at 1 week | 1 week
Time between pre-operative consultation and immediate information recall questionnaire | 24 hours
Time between pre-operative consultation and delayed information recall questionnaire | 1 week
Educational level | 30 months
Cognitive functioning | 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessels RP. Patients' memory for medical information. J R Soc Med. 2003 May;96(5):219-22. doi: 10.1177/014107680309600504. No abstract available. PMID 12724430
- [Background] Rutten LJ, Arora NK, Bakos AD, Aziz N, Rowland J. Information needs and sources of information among cancer patients: a systematic review of research (1980-2003). Patient Educ Couns. 2005 Jun;57(3):250-61. doi: 10.1016/j.pec.2004.06.006. PMID 15893206
- [Background] Watson PW, McKinstry B. A systematic review of interventions to improve recall of medical advice in healthcare consultations. J R Soc Med. 2009 Jun;102(6):235-43. doi: 10.1258/jrsm.2009.090013. PMID 19531618
- [Background] Phelps EE, Wellings R, Griffiths F, Hutchinson C, Kunar M. Do medical images aid understanding and recall of medical information? An experimental study comparing the experience of viewing no image, a 2D medical image and a 3D medical image alongside a diagnosis. Patient Educ Couns. 2017 Jun;100(6):1120-1127. doi: 10.1016/j.pec.2016.12.034. Epub 2016 Dec 30. PMID 28081938
- [Background] Zhuang YD, Zhou MC, Liu SC, Wu JF, Wang R, Chen CM. Effectiveness of personalized 3D printed models for patient education in degenerative lumbar disease. Patient Educ Couns. 2019 Oct;102(10):1875-1881. doi: 10.1016/j.pec.2019.05.006. Epub 2019 May 8. PMID 31113688
- [Background] van de Belt TH, Nijmeijer H, Grim D, Engelen LJLPG, Vreeken R, van Gelder MMHJ, Ter Laan M. Patient-Specific Actual-Size Three-Dimensional Printed Models for Patient Education in Glioma Treatment: First Experiences. World Neurosurg. 2018 Sep;117:e99-e105. doi: 10.1016/j.wneu.2018.05.190. Epub 2018 Jun 2. PMID 29870846
- [Background] Sezer S, Piai V, Kessels RPC, Ter Laan M. Information Recall in Pre-Operative Consultation for Glioma Surgery Using Actual Size Three-Dimensional Models. J Clin Med. 2020 Nov 13;9(11):3660. doi: 10.3390/jcm9113660. PMID 33203047